CLINICAL TRIAL: NCT02271958
Title: Mifepristone 2.5, 5, 10 mg Versus Placebo in the Treatment of Endometriosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mediterranea Medica S. L. (Other)
Responsible Party: Principal Investigator, Dr. Josep Lluis Carbonell i Esteve, Medical Director, Mediterranea Medica S. L.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Endomife 2,5/5/10/placebo
Record Dates: First submitted 2014-09-04; First posted 2014-10-22 (Estimated); Last update posted 2014-10-22 (Estimated); Status verified 2014-10

CONDITIONS: Endometriosis
Keywords: Mifepristone; Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Mifepristone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Experimental): Oral administration of 2,5 mg of mifepristone daily for 6 months
  Interventions: Drug: Mifepristone
- Group 2 (Experimental): Oral administration of 5 mg of mifepristone daily for 6 months
  Interventions: Drug: Mifepristone
- Group 3 (Experimental): Oral administration of 10 mg of mifepristone daily for 6 months
  Interventions: Drug: Mifepristone
- Group 4 (Experimental): Oral administration of mifepristone placebo daily for 3 months
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: Mifepristone
  Arms: Group 1; Group 2; Group 3
Drug: PLACEBO
  Arms: Group 4

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of 2.5, 5 and 10 mg doses of mifepristone against a placebo in women with laparoscopic diagnostic of endometriosis.

The hypothesis of the study is that the 5 mg mifepristone dose is safe and effective and should be used in future studies on medical treatment of endometriosis.

DETAILED DESCRIPTION:
This is double-blind randomized clinical trial.

Examinations undertaken Thorough gynecological examination, pelvic ultrasound examination, diagnostic laparoscopy before starting treatment in order to determine the localization, extent and degree of severity of the endometrial lesions and a score was assigned in accordance with the revised American Fertility Society (AFS) classification.19 Blood samples were taken for hematological tests and hepatic function. Endometrial biopsy was performed if endometrial thickness as calibrated by ultrasound was >8 mm or if there had been abnormal bleeding in the past 3 months. After 90 and 180 days of treatment an ultrasound examination of the pelvis was carried out and then followed by diagnostic-therapeutic laparoscopy and endometrial biopsy.

Subjects Women with laparoscopic confirmed diagnosis of endometriosis who volunteered to take part in the study. Inclusion criteria: a) age between 18 and 45, b) certain diagnosis of endometriosis of any degree corresponding to the American Fertility Society (AFS); c) patients with symptoms of endometriosis: dysmenorrhea or pelvic pain not attributable to other gynecological illness and d) acceptance of the use of barrier contraceptive methods during the study. Exclusion criteria: a) breastfeeding, b) hormonal or surgical treatment for the endometriosis less than 4 months previous to study, c) diabetes, d) severe arterial hypertension, e) hepatopathy, f) renal malfunction, g) endocrinopathy, and f) any other contraindication regarding the use of antiprogestins.

ELIGIBILITY:
Inclusion Criteria:

* Women with laparoscopic confirmed diagnosis of endometriosis
* Age between 18 and 45
* Certain diagnosis of endometriosis of any degree corresponding to the American Fertility Society (AFS)
* Patients with symptoms of endometriosis: dysmenorrhea or pelvic pain not attributable to other gynecological illness and
* Acceptance of the use of barrier contraceptive methods during the study

Exclusion Criteria:

* Breastfeeding
* Hormonal or surgical treatment for the endometriosis less than 4 months previous to study
* Diabetes
* Severe arterial hypertension
* Hepatopathy
* Renal malfunction
* Endocrinopathy
* Any other contraindication regarding the use of antiprogestins.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 360 (Actual)
Dates: Start 2010-11; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Changes in prevalence of dysmenorrhea and the average reduction in its intensity. | 6 months
  The principal variables in evaluating effectiveness were the percentage changes in prevalence of dysmenorrhea and the average reduction in its intensity.
Incidence of hot flushes, nausea, dizzy spells, vomiting, fatigue/tiredness, raised hepatic transaminases, histological alterations of the endometrium. | 6 months
  Safety was evaluated by the incidence of hot flushes, nausea, dizzy spells, vomiting, fatigue/tiredness, raised hepatic transaminases, histological alterations of the endometrium.
Changes in scores according to American Fertility Society (AFS) | 6 months
  Effectiveness was assessed by measuring changes in scores according to American Fertility Society (AFS)

CONTACTS AND LOCATIONS:
Overall Officials: Josep Ll Carbonell, Doctor, Principal Investigator — Medical Clinic Mediterranea
Locations (1):
- Hospital Eusebio Hernández, "Maternidad Obrera", Havana, La Habana, Cuba

REFERENCES:
- [Derived] Chen I, Kives S, Zakhari A, Nguyen DB, Goldberg HR, Choudhry AJ, Le AL, Kowalczewski E, Schroll JB. Progestagens for pain symptoms associated with endometriosis. Cochrane Database Syst Rev. 2025 Oct 9;10(10):CD002122. doi: 10.1002/14651858.CD002122.pub3. PMID 41065045